CLINICAL TRIAL: NCT05359237
Title: A Pharmacokinetic Study of VinCRIStine in Infants Dosed According to BSA-Banded Infant Dosing Tables and Older Children Dosed by Traditional BSA Methods
Brief Title: Vincristine Pharmacokinetics in Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PEPN22P1; NCI-2022-03576 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN22P1 (Other: Pediatric Early Phase Clinical Trial Network); PEPN22P1 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Specimen Handling; Vincristine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (SOC vincristine, biospecimen collection): Patients receive vincristine IV per SOC. Patients undergo collection of blood samples at baseline (before first vincristine dose), and 2, 6-8, and 18-24 hours after a dose of vincristine. Patients may also undergo collection of blood samples with a second SOC vincristine dose at the same time points.
  Interventions: Procedure: Biospecimen Collection; Drug: Vincristine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Vincristine — Given IV per standard of care
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This pilot trial compares drug exposure levels using a new method for dosing vincristine in infants and young children compared to the standard dosing method based on body surface area (BSA) in older children. Vincristine is an anticancer drug used to a variety of childhood cancers. The doses anticancer drugs in children must be adjusted based on the size of the child because children vary significantly in size (height, weight, and BSA) and ability to metabolize drugs from infancy to adolescence. The dose of most anticancer drugs is adjusted to BSA, which is calculated from a patient's weight and height. However, infants and young children have more severe side effects if the BSA is used to calculate their dose, so new dosing models have to be made to safely give anticancer drugs to the youngest patients. This new method uses a BSA-banded approach to determine the dose. Collecting blood samples before and after a dose of the drug will help researchers determine whether this new vincristine dosing method results in equivalent drug levels in the blood over time in infants and young children compared to older children.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To validate body surface area (BSA)-banded infant dosing tables by comparing vinCRIStine drug exposure, defined as the area under the concentration-time curve for the elimination phase (AUCelim), in infants and young children dosed according to the table to older children dosed according to BSA.

SECONDARY OBJECTIVE:

I. To estimate intra- and inter-age group variability (CV) using non-compartmental analysis (NCA) and population pharmacokinetic (PK) methods.

EXPLORATORY OBJECTIVES:

I. To correlate higher AUCelim with the presence of functionally impaired single nucleotide polymorphisms (SNP) of CYP3A4 and CYP3A5.

II. To assess vinCRIStine dose modifications in infants receiving weekly vinCRIStine dosed according to the BSA-banded infant dosing tables.

OUTLINE:

Patients receive vincristine intravenously (IV) per standard of care (SOC). Patients undergo collection of blood samples at baseline (before first vincristine dose), and 2, 6-8, and 18-24 hours after a dose of vincristine. Patients may also undergo collection of blood samples with a second SOC vincristine dose at the same time points.

Patients are followed for dose modifications for a period of 42 days (when receiving weekly dosing of vincristine).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be =< 12 years of age at the time of study enrollment. Patients will be stratified into 4 age groups:

  * 0 to 6 months
  * 6 months and 1 day to 12 months
  * 12 months and 1 day to 36 months
  * 36 months and 1 day to 12 years with a BSA ≥ 0.6 m^2
* Newly diagnosed and relapsed cancer diagnosis that is being treated with vinCRIStine at the 1.5 mg/m^2 dose level
* Any disease status
* Patients must have a Lansky performance status of 50 or higher
* Patients must be receiving a treatment regimen that includes 1.5 mg/m^2 vinCRIStine (maximum dose 2 mg)
* Patients with a BSA < 0.6 m^2 must be dosed according to the Children's Oncology Group (COG) BSA-banded infant dosing table for the 1.5mg/m2 dose level for vinCRIStine

  * Note: Patients can be studied after any dose of vinCRIStine
* Patients who are NOT enrolled on a COG clinical trial and who have a BSA < 0.6 m^2 and who are being dosed according to another infant dosing method (e.g., the 30-Rule) can receive a dose of vinCRIStine from the infant dosing table for the pharmacokinetic study. These patients will NOT be part of the Dose Modification Assessment
* Patients with a seizure disorder may be enrolled if on allowable anticonvulsants and well controlled as evidenced by no increase in seizure frequency in the prior 7 days
* Nervous system toxicities (Common Terminology Criteria for Adverse Events [CTCAE]) version (v)5 resulting from prior therapy must be grade =< 2
* Central venous access device in place (e.g., percutaneous indwelling central catheter [PICC], port, Broviac) or scheduled to be placed prior to the dose of vinCRIStine and that can be used for pharmacokinetic (PK) sampling
* VinCRIStine may be given as an outpatient, as long as all sample time points can be collected, which will require return for hour 24 sampling

Exclusion Criteria:

* Azoles antifungals and macrolide antibiotics: Patients who are currently receiving an azole or macrolide (e.g., fluconazole, isavuconazole, itraconazole, posaconazole, voriconazole, ketoconazole, eryromycin, clarithromycin, azithromycin, roxithromycin, or telithromycin) are not eligible
* CYP3A4/5 inducers/inhibitors: Patients receiving any medications or substances that are considered moderate or strong inhibitors or inducers of CYP3A4/5 are not eligible. Moderate or strong inducers or inhibitors of CYP3A4/5 should be avoided from 14 days prior to enrollment to the end of the study.

  * Note the following are allowed:

    * Dexamethasone for CNS tumors or metastases, on a stable dose
    * Aprepitant for management of nausea and vomiting
* Anticonvulsants: Patients receiving moderate or strong CYP3A4/5 enzyme inducing anticonvulsants are not eligible.
* Patients with Charcot-Marie-Tooth disease
* A baseline neurological disorder with manifestations that overlap with vinCRIStine-associated neurotoxicities
* Patients being treated on a Children Oncology Group (COG) clinical trial, that does not use the infant dosing tables for vinCRIStine are not eligible for this study.
* Patients receiving a modified dose (< 1.5 mg/m^2) of vinCRIStine due to prior toxicity
* Patients who in the opinion of the investigator may not be able to comply with the sampling requirements of the study

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and young children receiving treatment regimen that includes vinCRIStine
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration time curve for the elimination phase (AUCelim) by age group | Up to 24 hours post vincristine dose
  Estimate (95% CI) of the mean area under the concentration time curve for the elimination phase assessed at 0, 2, 6-8, and 18-24 hours after vinCRISTine dose by age group.

SECONDARY OUTCOMES:
Intra- and inter-age coefficient of variation (CV) | Up to 42 days
  Estimate of the intra- and inter-age coefficient of variation using non-compartmental analysis (NCA) and population pharmacokinetic (PK) methods.

OTHER OUTCOMES:
Correlation of AUC for the elimination phase with CYP3A4 and CYP3A5 single nucleotide polymorphisms (SNPs) | Up to 24 hours
  Correlate AUCelim with the presence of functionally impaired single nucleotide polymorphisms (SNP) of CYP3A4 and CYP3A5.
Number of patients requiring vincristine dose modifications | Up to 42 days
  Number of patients requiring vincristine dose modifications stratified by age group.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Blauel, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (29):
- United States (27):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Queensland Children's Hospital, South Brisbane, Queensland, Australia
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada